CLINICAL TRIAL: NCT01569672
Title: Ohio Patient Navigation Research Program
Brief Title: Ohio Patient Navigator Research Program
Acronym: OPNRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OPNRP; SIRG-05-253-01 (Other Grant/Funding Number: American Cancer Society); NCI-2012-00205 (Registry Identifier: Clinical Trials Reporting Program (CTRP)); OSU-6100 (Other: OSU)
Record Dates: First submitted 2012-03-19; First posted 2012-04-03 (Estimated); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer; Cervical Cancer; Colon Cancer; Rectal Cancer; Abnormal Breast Cancer Screening Tests; Abnormal Cervical Cancer Screening Tests; Abnormal Colon Cancer Screening Tests
Keywords: Navigator
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Clinic (Active Comparator): Patient Navigator matched with subjects. Patient Navigators will be matched with subjects at the intervention clinics and will assist patients with questions, issues or concerns with their cancer treatment/diagnosis or abnormal test results and followup test or treatments
  Interventions: Behavioral: Patient Navigator matched with subject
- Control Clinics (Placebo Comparator): Subjects are mailed informational/educational materials.
  Interventions: Behavioral: Subjects are mailed informational/educational materials

INTERVENTIONS:
Behavioral: Patient Navigator matched with subject — Subject is matched with a patient navigator. The patient navigator calls the patient. The amount of time between the abnormal test and treatment will be measured.
  Arms: Intervention Clinic
Behavioral: Subjects are mailed informational/educational materials — Subjects will be mailed informational/educational materials. The amount of time between the abnormal test and treatment will be measured.
  Arms: Control Clinics

SUMMARY:
The Ohio Patient Navigator Research Program (OPNRP) proposes to alleviate disparities in relation to the timely diagnosis and treatment of breast, cervical and colorectal cancer in Columbus, OH.

DETAILED DESCRIPTION:
The goal of the Ohio Patient Navigator Research Program (OPNRP) is to facilitate timely access to quality, standard cancer care for persons diagnosed with breast, cervical, and colorectal cancer in a culturally sensitive manner. This program will be carried out within clinics of The Ohio State University Primary Care Network (OSU PCN) and the Columbus Neighborhood Health Centers (CNHC) in Columbus, Ohio with a preponderance of patients from underserved (i.e., racial/ethnic minorities, people of lower socioeconomic status, and the elderly) populations. This goal will be accomplished by completing the following objectives:

Objectives

* Develop the OPNRP through the work of a consortium of institutions including The Ohio State University Comprehensive Cancer Center (OSUCCC) and James Cancer Hospital (JCH), the Ohio Division of the American Cancer Society (ACS), and the Ohio Commission on Minority Health (OCMH);
* Conduct a formative research phase to assess referral patterns and barriers to prompt diagnosis and treatment services, as well as strategies to overcome barriers among patients of these clinic networks;
* Implement and evaluate the patient navigator program in 12 primary care clinics using a group randomized, controlled design to assess the efficacy of the intervention to reduce the time to delivery of standard cancer diagnosis and services and non-cancer resolution or cancer diagnosis and treatment after the diagnosis of an abnormal finding from a cancer detection procedure for breast, cervical or colorectal cancer, as well as improve patient satisfaction with care and quality of life;
* Conduct a process evaluation to assess the barriers to implementation of the intervention program, the features of the intervention (e.g., appointments kept/missed, materials provided to patients, etc.), patient satisfaction with the navigator, and clinic perceptions of the navigator program; and
* Conduct a cost-effectiveness evaluation of the navigator program. Results from this study will be disseminated throughout Ohio by community partners and used to provide information on concrete ways to utilize patient navigators to reduce the burden of cancer in underserved populations, a goal of the National Cancer Institute (NCI) and Department of Health and Human Services (DHS) Healthy People 2010. The OPNRP is one of nine grantees in NCI/ACS's Patient Navigator Research Program (PNRP).

ELIGIBILITY:
Inclusion Criteria:

* Over age 18 years
* Be a regular patient of the primary care practice
* Be able to give informed consent
* Have had either an abnormal screening test, an abnormal diagnostic test, or an abnormal clinical finding leading to diagnostic testing for cervical, breast, or colorectal cancer, or a diagnosis of cervical, breast, or colorectal cancer
* Speak and understand English, or Spanish. For those participants who do not speak and understand English they will only be enrolled/consented into the program if translation services are available.

Exclusion Criteria:

* Cognitively impaired
* Prior history of cancer (except for nonmelanoma of the skin)
* Living in a nursing home
* Prior navigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 941 (Actual)
Dates: Start 2006-11; Primary Completion 2010-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Amount of time from abnormal evaluation of the breast, cervix, and colon or rectum to needed tests and treatment | Up to one year
  How much time exist between an abnormal test diagnosis for breast, cervical or colon or rectum cancer to when the needed follow up tests or treatment is done.

SECONDARY OUTCOMES:
Number of barriers and effect of barriers on receiving needed tests and treatment | 1 year
  List of and number of barriers and qualitatively how they influence a person's reasons for not getting a needed screening test or treatment

CONTACTS AND LOCATIONS:
Overall Officials: Electra D Paskett, PhD, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (1):
- The Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Battaglia TA, Darnell JS, Ko N, Snyder F, Paskett ED, Wells KJ, Whitley EM, Griggs JJ, Karnad A, Young H, Warren-Mears V, Simon MA, Calhoun E. The impact of patient navigation on the delivery of diagnostic breast cancer care in the National Patient Navigation Research Program: a prospective meta-analysis. Breast Cancer Res Treat. 2016 Aug;158(3):523-34. doi: 10.1007/s10549-016-3887-8. Epub 2016 Jul 18. PMID 27432417
- [Derived] Wells KJ, Winters PC, Jean-Pierre P, Warren-Mears V, Post D, Van Duyn MA, Fiscella K, Darnell J, Freund KM; Patient Navigation Research Program Investigators. Effect of patient navigation on satisfaction with cancer-related care. Support Care Cancer. 2016 Apr;24(4):1729-53. doi: 10.1007/s00520-015-2946-8. Epub 2015 Oct 5. PMID 26438146
- [Derived] Rodday AM, Parsons SK, Snyder F, Simon MA, Llanos AA, Warren-Mears V, Dudley D, Lee JH, Patierno SR, Markossian TW, Sanders M, Whitley EM, Freund KM. Impact of patient navigation in eliminating economic disparities in cancer care. Cancer. 2015 Nov 15;121(22):4025-34. doi: 10.1002/cncr.29612. Epub 2015 Sep 8. PMID 26348120
- [Derived] Ko NY, Darnell JS, Calhoun E, Freund KM, Wells KJ, Shapiro CL, Dudley DJ, Patierno SR, Fiscella K, Raich P, Battaglia TA. Can patient navigation improve receipt of recommended breast cancer care? Evidence from the National Patient Navigation Research Program. J Clin Oncol. 2014 Sep 1;32(25):2758-64. doi: 10.1200/JCO.2013.53.6037. Epub 2014 Jul 28. PMID 25071111
- See also: Jamesline — http://cancer.osu.edu